CLINICAL TRIAL: NCT01550510
Title: Phase I/II Study of Intravenous Ascorbic Acid in Combination With Irinotecan Versus Irinotecan Alone for Advanced Colorectal Cancer
Brief Title: Research Study of IV Vitamin C in Combination With Irinotecan vs Irinotecan Alone for Advanced Colorectal CA
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Closed: low enrollment, many treatment options available for Colorectal Cancer
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11D.459; JT 1548 (Other: JeffTrial Number)
Record Dates: First submitted 2012-02-23; First posted 2012-03-12 (Estimated); Results first posted 2018-08-24 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Stage IV Colorectal Cancer
Keywords: Stage IV Colorectal cancer; Colorectal Neoplasms; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Neoplasms; Digestive System Diseases; Gastrointestinal Diseases; Colonic Diseases; Intestinal Diseases; Rectal Diseases; Ascorbic Acid; Vitamins; Irinotecan; Integrative Medicine; Complementary Medicine; Alternative Medicine Antioxidants; Molecular Mechanisms of Pharmacological Action; Pharmacologic Actions; Protective Agents; Physiological Effects of Drugs; Micronutrients; Growth Substances; Antineoplastic Agents, Phytogenic; Antineoplastic Agents; Therapeutic Uses; Radiation-Sensitizing Agents; Topoisomerase I Inhibitors; Topoisomerase Inhibitors; Enzyme Inhibitors
MeSH Terms: conditions — Colorectal Neoplasms; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Neoplasms; Digestive System Diseases; Gastrointestinal Diseases; Colonic Diseases; Intestinal Diseases; Rectal Diseases | interventions — Ascorbic Acid; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ascorbic Acid + Irinotecan (Experimental): Ascorbic Acid (50-100g, 3x weekly) with 350mg/m2 irinotecan once a week every 3 weeks
  Interventions: Drug: Ascorbic Acid; Drug: Irinotecan
- Standard of Care (irinotecan alone) (Active Comparator): 350mg/m2 irinotecan once a week every 3 weeks
  Interventions: Drug: Irinotecan

INTERVENTIONS:
Drug: Ascorbic Acid — 3x a week for 9 weeks
  Other Names: Ascorbate; Vitamin C
  Arms: Ascorbic Acid + Irinotecan
Drug: Irinotecan — 350mg/m2 once a week every 3 weeks
  Other Names: Camptothecin-11; CPT-11

SUMMARY:
This protocol is a phase I/II, study of ascorbic acid (AA) infusions combined with treatment with irinotecan versus treatment with irinotecan alone in patients with recurrent or advanced colorectal cancer who have failed at least one treatment regimen with a 5-FU based therapy. This study will be conducted as an amendment to Investigational New Drug # 77486.

DETAILED DESCRIPTION:
Phase I: To assess whether or not (IV) Ascorbic Acid (AA) with irinotecan therapy is relatively safe and well-tolerated. This aim will be assessed by enrolling a minimum of 6 subjects meeting inclusion criteria, using a modified 3+3 design. Safety will be assessed with the following: toxicity graded by the NCI CTC, urinalysis pre- and post-infusion, basic metabolic panel, and CBC. From our experience and in the experience of our study collaborators, we hypothesize that the combination of IV AA with irinotecan will not be associated with adverse events.

Phase II: To utilize CT or PET/CT (when available) scans to evaluate disease progression to assess overall tumor response rate (complete and partial response) in subjects with advanced or recurrent colorectal cancer treated with the combination of ascorbic acid and irinotecan versus irinotecan alone.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Metastatic colorectal carcinoma (stage IV disease).
* Patients must have progressed on one or more prior chemotherapy treatment regimens including at least one trial of a 5-FU/oxaliplatin based therapy (FOLFOX) in combination with bevacizumab. Patients must not have had standard chemotherapy within at least 2 weeks of beginning ascorbic acid treatment provided that they have recovered from any toxicities that they experienced.
* G6PD status > lower limit of normal
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2.
* Laboratory at baseline evaluation for inclusion in the study: creatinine ≤1.5X upper limit (if the creatinine is elevated, but ≤1.5X the ULN, a 24 hour creatinine clearance will be obtained); transaminase (AST/ALT) ≤2.0X upper limit of normal; bilirubin levels ≥ 2 mg/dL; ANC ≥1,500/mm3; Hemoglobin > 8g/dL; platelet ≥ 100,000/mm3;
* Women of childbearing potential will confirm a negative pregnancy test and must practice effective contraception during the study.
* Willing and able to provide informed consent and participate in the study procedures.

Exclusion Criteria:

* Patients with evidence of a significant current psychiatric disorder that would prevent completion of the study as determined by the PI will not be allowed to participate.
* Co-morbid medical condition that would affect survival or tolerance as determined by the PI. This includes patients who have not fully recovered from toxicities associated with prior therapy. It also includes subjects who, as determined by the PI, are at risk of experiencing fluid overload (i.e., congestive heart failure).
* Patients who currently abuse alcohol or drugs.
* Patients with known glomerular filtration rate of <60ml/min or with nephrotic range proteinuria.
* Pregnant or lactating women
* Enrollment in active clinical trial/ experimental therapy or IND study within the prior 30 days.
* Contraindication for CT or PET/CT as per the PI.
* Patients who are on strong inducers of CYP3A4 which include but are not limited to: Aminoglutethimide, Bexarotene, Bosentan, Carbamazepine, Dexamethasone, Efavirenz, Fosphenytoin, Griseofulvin, Modafinil, Nafcillin, Nevirapine, Oxcarbazepine, Phenobarbital, Phenytoin, Primidone, Rifabutin, Rifampin, Rifapentine, St. John's wort.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-12; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A Monti, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/

RESULTS

PARTICIPANT FLOW:
Groups:
- Ascorbic Acid: Ascorbic Acid (50-100g, 3x weekly)
  Ascorbic Acid: 3x a week for 9 weeks
- Standard of Care (Irinotecan Alone): 350mg/m2 once a week every 3 weeks
Period: Overall Study
Arm/Group | Ascorbic Acid | Standard of Care (Irinotecan Alone)
Started | 4 | 0
Completed | 4 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Phase 2 portion of this study never enrolled and therefore no patients were enrolled to the standard of care arm.
Groups:
- Ascorbic Acid+Irinotecan: Ascorbic Acid (50-100g, 3x weekly)
  Ascorbic Acid: 3x a week for 9 weeks
- Total: Total of all reporting groups
Arm/Group | Ascorbic Acid+Irinotecan | Standard of Care (Irinotecan Alone) | Total
Number analyzed (Participants) | 4 | 0 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 1 |  | 1
  >=65 years | 3 |  | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 |  | 3
  Male | 1 |  | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 4 |  | 4
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 2 |  | 2
  White | 1 |  | 1
  More than one race | 0 |  | 0
  Unknown or Not Reported | 1 |  | 1
Region of Enrollment [Number; unit: participants]
  United States | 4 |  | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Experience Serious Adverse Events as Defined by the Common Terminology Criteria for Adverse Events (CTCAE) v4.0.
Description: Safety: The primary aim is to assess whether or not (IV) Ascorbic Acid (AA) with irinotecan therapy is relatively safe and well-tolerated according to Common Terminology Criteria for Adverse Events (CTCAE) v4.0.
Time Frame: 9 weeks +/- 2 weeks
Population: The study was closed early due to lack of accrual. The data were not collected or analyzed.
Arm/Group | Ascorbic Acid+Irinotecan | Standard of Care (Irinotecan Alone)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number of Participants That Are Alive After 11 Weeks.
Description: To evaluate progression-free survival related to treatment of patients with advanced or recurrent colorectal cancer
Time Frame: 9 weeks +/- 2 weeks
Population: The study was closed early due to lack of accrual. The data were not collected or analyzed.
Arm/Group | Ascorbic Acid | Standard of Care (Irinotecan Alone)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The study was closed early due to lack of accrual. Adverse event data were collected for the patients who were enrolled in the study.
Arm/Group | Ascorbic Acid+Irinotecan | Standard of Care (Irinotecan Alone)
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/0
Other Adverse Events (participants affected / at risk) | 2/4 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ascorbic Acid+Irinotecan (N=4) | Standard of Care (Irinotecan Alone) (N=0)
Hypokalemia (Blood and lymphatic system disorders) | 1 (1) | NA
Low Hemoglobin (Blood and lymphatic system disorders) | 1 (1) | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes